CLINICAL TRIAL: NCT06457386
Title: Echocardiography Versus no Echocardiography in Individuals With Staphylococcus Aureus Bacteremia and a VIRSTA Score <3: a Non-inferiority Randomized Controlled Trial
Brief Title: Echocardiography Versus no Echocardiography in S. Aureus Bacteraemia and VIRSTA Score < 3
Acronym: VIRSTA-VAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: APHP220807; 2023-A01572-43 (Other: ID-RCB)
Record Dates: First submitted 2024-06-03; First posted 2024-06-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Staphylococcus Aureus; Bacteremia; Infective Endocarditis
Keywords: VIRSTA score < 3; Staphylococcus aureus bacteraemia; Echocardiography; Infective endocarditis
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia; Endocarditis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systematic echocardiography arm (Active Comparator): "transthoracic echocardiography (TTE) will be performed as soon as possible within 14 days following the first blood sample collection for SAB diagnosis, completed, if required, by a transoesophageal (TEE) echocardiography based on the judgment of the echocardiographist.
  SAB in patients of both arms will be treated according to current recommendations, taking into account the result of the echocardiography in the control arm. "
  Interventions: Procedure: systematic echocardiography
- no echocardiography arm (Experimental): "no echocardiography will be performed unless occurrence of new events evocating IE (extra-cardiac events or positive Staphylococcus aureus blood culture), based on the clinical judgment of the investigator.
  SAB in patients of both arms will be treated according to current recommendations, taking into account the result of the echocardiography in the control arm.
  "
  Interventions: Procedure: no echocardiography arm

INTERVENTIONS:
Procedure: systematic echocardiography — "transthoracic echocardiography (TTE) will be performed as soon as possible within 14 days following the first blood sample collection for SAB diagnosis, completed, if required, by a transoesophageal (TEE) echocardiography based on the judgment of the echocardiographist.
  SAB in patients of both arms will be treated according to current recommendations, taking into account the result of the echocardiography in the control arm. "
  Arms: systematic echocardiography arm
Procedure: no echocardiography arm — "no echocardiography will be performed unless occurrence of new events evocating IE (extra-cardiac events or positive Staphylococcus aureus blood culture), based on the clinical judgment of the investigator.
  SAB in patients of both arms will be treated according to current recommendations, taking into account the result of the echocardiography in the control arm. "
  Arms: no echocardiography arm

SUMMARY:
Staphylococcus aureus is the most frequent cause of both healthcare-associated and community-acquired bloodstream infections worldwide. Infective endocarditis (IE) has been detected in 5-17% of cases and is a determinant of poor prognosis. The investigators developed a score (the VIRSTA score) based on patients' characteristics to rule out IE with high confidence (negative predictive value (NPV) above 99%) in patients with SAB. This score, with a cut-off of 3 has been externally validated by two international studies which have also established its high NPV. The 2023 European society of cardiology (ESC) guidelines state that echocardiography should be considered in all patients with Staphylococcus aureus bacteremia (SAB) using risk scores (including VIRSTA score) to guide the use or not of echocardiography. While recommended, the investigators think that VIRSTA score must be evaluated in terms of patients' outcome.

DETAILED DESCRIPTION:
In the interventional arm (no-echocardiography strategy) without echocardiography, at the individual level, not performing an echocardiography will avoid a useless examination, the mobilization of the patient and the discomfort related to its performance.

In this arm, the theoretical risk is to diagnose Infective endocarditis (IE ) only at a later phase stage, i.e., at a phase of symptomatic manifestation of valve regurgitation or at the occurrence of relapse of bacteremia due to insufficient duration of antibiotic treatment. It should be noted that patients with prosthetic valve, who have "de facto" a VIRSTA score > 3, will therefore not be included in the protocol. Given the expected rarity of IE in patients with a VIRSTA score <3 and the theoretical consequences of not performing echocardiography, the primary endpoint chosen will be mortality and Staphylococcus aureus bacteraemia (SAB) relapse. The endpoint will be assessed at 90 days and not at discharge to capture relapses of inadequately treated bacteremia and the mid-term consequences of a possible delay in IE diagnosis.

On a collective scale, not performing echocardiography in many patients in whom it is not useful will allow resources to be allocated to the individuals who need it most.

ELIGIBILITY:
Inclusion criteria

* Volunteers over 18 years of age;
* Hospitalized with at least one blood culture positive for Staphylococcus aureus;
* At the time of inclusion, negative control blood culture performed 48 hours after the first Staphylococcus aureus blood culture collection;
* VIRSTA score < 3; Exclusion criteria
* Patient with catheter colonization without SAB, defined as positive blood cultures only through vascular access device specimen;
* Patient referred to the hospital for the management of IE;
* Contra indication to transthoracic echocardiography (TTE);
* Echocardiography already performed before inclusion (TTE or TEE) for the current SAB;
* Pregnancy;
* Patient under guardianship or trusteeship.
* Absence of written informed consent from the patient
* No affiliation to social security (beneficiary or assignee)
* Subject already involved in another interventional clinical research for which echocardiography must be done"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
All causes mortality | 90 Days
SAB relapse microbiologically confirmed | 90 Days
  Relapse of SAB is defined in patients with bacteriologic success as the isolation of a strain of Staphylococcus aureus with in vitro antibiotic susceptibility pattern similar to that of the Staphylococcus aureus strain isolated at inclusion. Relapse will be confirmed at the end of the study by an independent adjudication committee

SECONDARY OUTCOMES:
Number of definite IE according to ESC 2023 criteria | the end of hospital stay, up to 90 days
  An independent adjudication committee will classify definite, possible or excluded IE according to the 2023 ESC criteria
Number of definite IE according to ESC 2023 criteria | 90 Days
Number of IE valvular cardiac surgery and indications (heart failure, uncontrolled infection or prevention of embolism) | the end of hospital stay, up to 90 days
Number of IE valvular cardiac surgery and indications (heart failure, uncontrolled infection or prevention of embolism) | 90 Days
Length of hospitalization (days) | 180 Days
All-causes mortality | 180 Days
Number of SAB relapse | 90 Days
Cost difference between the two strategies | 90 Days
  Cost-effectiveness analysis if there is a difference in the number of events in each arm
quality of life measured by EQ5D5L | 180 Days

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Duval, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bichat Claude Bernard Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided